CLINICAL TRIAL: NCT07325539
Title: Low-dose Radiotherapy (LDRT) Combined With Toripalimab and GP Chemotherapy for Recurrent/Metastatic Nasopharyngeal Carcinoma (LIGHT): A Single-Center, Open-Label, Single-Arm Phase II Clinical Study
Brief Title: LDRT Combined With Toripalimab and Chemotherapy for Recurrent/Metastatic NPC
Acronym: LIGHT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-451-FLK
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Nasopharyngeal Cancinoma (NPC); Nasopharangeal Cancer
Keywords: PD-1 antibody; Low dose radiotherapy; Recurrent/Metastatic Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDRT + Toripalimab + GP chemotherapy (Experimental): Patients will receive LDRT plus toripalimab and GP chemotherapy for 4-6 cycles, then followed by toripalimab until disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine(GEM); Drug: Cisplatin; Drug: Toripalimab; Radiation: LDRT

INTERVENTIONS:
Drug: Gemcitabine(GEM) — Gemcitabine 1000mg/m2, d1 & 8 of every cycle, every 3 weeks for 4-6 cycles
Drug: Cisplatin — Cisplatin 80mg/m2, d1 of every cycle, every 3 weeks for 4-6 cycles
Drug: Toripalimab — Toripalimab 240 mg, d1of every cycle, every 3 weeks for 4-6 cycles. Toripalimab maintenance, 240 mg, d1of every cycle, every 3 weeks until disease progression or unacceptable toxicity.
Radiation: LDRT — Irradiation of the primary lesion and regional metastatic lymph nodes, 0.5 Gy per fraction for 4 fractions, d0-3, every 3 weeks for 4-6 cycles

SUMMARY:
This study aims to evaluate the efficacy and safety of LDRT combined with toripalimab and GP chemotherapy in patients with recurrent or metastatic nasopharyngeal carcinoma through a prospective, open-label, single-arm Phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old.
* Histologically confirmed non-keratinizing nasopharyngeal carcinoma (WHO Type II or III).
* ECOG Performance Status score of 0-1.
* At least one measurable lesion as per RECIST v1.1 criteria.
* Patients with newly diagnosed metastatic NPC, or patients with locoregionally advanced NPC who developed metastasis ≥6 months or recurrence ≥12 months after completing radical radiotherapy/chemotherapy for the primary lesion.
* No prior radiotherapy, chemotherapy, immunotherapy, or biological therapy for recurrent/metastatic lesions.
* Adequate organ function, meeting the following criteria within 7 days prior to treatment:

  1. Hematological criteria (without transfusion or hematopoietic growth factor support within 14 days):

     1. Hemoglobin (Hb) ≥90 g/L.
     2. White Blood Cell (WBC) count ≥4.0 × 10⁹/L.
     3. Platelet count (PLT) ≥100 × 10⁹/L.
  2. Biochemical criteria:

     1. Total Bilirubin (TBIL) ≤1.5 × Upper Limit of Normal (ULN).
     2. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤2.5 × ULN.
     3. Serum Creatinine (Cr) ≤1.5 × ULN AND Creatinine Clearance (CCr) ≥60 mL/min.
  3. Coagulation function: INR and APTT ≤1.5 × ULN.
  4. Normal results for myocardial injury markers, heart failure markers, and electrocardiogram (ECG). For patients with abnormal results in any of these, the investigator will assess the need for Doppler echocardiography.
  5. Thyroid function: TSH ≤ ULN. If abnormal, FT3 and FT4 levels should be considered; patients can be enrolled if FT3 and FT4 levels are normal.
* Women of childbearing potential must have used reliable contraception, have a negative serum pregnancy test within 7 days before enrollment, and be willing to use adequate contraception during the trial and for 8 weeks after the last dose of the study drug, or be surgically sterile. Men must agree to use adequate contraception or be surgically sterile during the trial and for 8 weeks after the last dose.
* Voluntary provision of signed informed consent, with good compliance.

Exclusion Criteria:

* Disease progression within 6 months after completing standard treatment for locoregionally advanced nasopharyngeal carcinoma.
* Absence of identifiable tumor lesions in both the primary site and locoregional lymph nodes, precluding the development of an LDRT plan.
* Inability to undergo MRI due to reasons such as implanted metal devices or claustrophobia.
* Requirement for systemic use of corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose or during the study. Inhaled or topical steroids and adrenal replacement steroid doses >10 mg/day prednisone equivalent are permitted in the absence of active autoimmune disease. Physiological replacement doses of corticosteroids (≤10 mg/day prednisone equivalent) are allowed.
* Recurrent target lesions suitable for curative surgery or a second course of radiotherapy.
* History of any active autoimmune or autoimmune disease, or known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation. Exceptions include type I diabetes, hypothyroidism requiring hormone replacement therapy, and skin disorders not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
* Active or uncontrolled severe infection (≥CTCAE Grade 3) within 4 weeks prior to enrollment.
* History of active tuberculosis within the past year, regardless of treatment. Patients with a history of active pulmonary tuberculosis over 1 year ago who have documented evidence of adequate past anti-tuberculosis treatment may be considered; otherwise, they are excluded.
* History of hypertension that cannot be adequately controlled with a single antihypertensive medication (systolic BP ≥150 mmHg or diastolic BP ≥90 mmHg).
* Clinically significant bleeding symptoms or definite bleeding tendency, specifically excluding cases of local recurrence with high bleeding risk or cases within 1 year post-radiotherapy assessed to have a high risk of necrosis.
* Urinalysis showing urine protein ≥ ++ AND confirmed 24-hour urine protein ≥1.0 g.
* Myocardial ischemia (above Grade I), myocardial infarction, arrhythmia (including QTc ≥480 ms), or ≥ Grade 2 congestive heart failure (NYHA classification) within 6 months prior to enrollment.
* If an echocardiogram is required per Inclusion Criterion 7(4), results showing Left Ventricular Ejection Fraction (LVEF) below the lower limit of normal (60%).
* Diagnosis of other malignancies within 5 years prior to enrollment, except for cured non-melanoma skin cancer, carcinoma in situ of the cervix, and papillary thyroid carcinoma.
* Presence of leptomeningeal or central nervous system metastases.
* HIV positive, TP positive, liver cirrhosis, decompensated liver disease, active hepatitis (uncontrolled active hepatitis despite treatment: Hepatitis B - HBsAg positive and HBV DNA ≥1 × 10⁴ copies/mL; Hepatitis C - HCV RNA positive with abnormal liver function; co-infection with HBV and HCV) requiring antiviral therapy.
* Participation in another anti-tumor drug clinical trial within 4 weeks prior to enrollment.
* Administration of any live attenuated vaccine within 30 days prior to enrollment.
* Contraindications to radiotherapy.
* Known allergy to the study drug or any of its excipients, or history of severe allergic reactions to other monoclonal antibodies.
* History of psychoactive drug abuse unable to be abstained, or presence of psychiatric disorders.
* Any other condition assessed by the investigator as potentially endangering the patient's safety or compliance, including severe concurrent diseases (including psychiatric disorders) requiring prompt treatment, severely abnormal laboratory test results, or other psychological, familial, or sociological factors deemed high-risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by RECIST 1.1 | up to approximately 2 years
  PFS was defined as the time from enrollment to the first occurrence of disease progression as determined according to RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | up to approximately 2 years
  The proportion of patients who achieved a complete response (CR) or partial response (PR), assessed according to RECIST v1.1.
Progression-free survival (PFS) assessed by iRECIST | up to approximately 2 years
  PFS was defined as the time from enrollment to the first occurrence of disease progression as determined according to iRECIST or death from any cause, whichever occurs first.
Overall survival (OS) | up to approximately 4 years
  OS was defined as the time from enrollment to death from any cause.
Adverse events | up to approximately 2 years
  All adverse event or serious adverse event that occurred during the study period according to CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee N, Harris J, Garden AS, Straube W, Glisson B, Xia P, Bosch W, Morrison WH, Quivey J, Thorstad W, Jones C, Ang KK. Intensity-modulated radiation therapy with or without chemotherapy for nasopharyngeal carcinoma: radiation therapy oncology group phase II trial 0225. J Clin Oncol. 2009 Aug 1;27(22):3684-90. doi: 10.1200/JCO.2008.19.9109. Epub 2009 Jun 29. PMID 19564532
- [Result] Lee NY, Zhang Q, Pfister DG, Kim J, Garden AS, Mechalakos J, Hu K, Le QT, Colevas AD, Glisson BS, Chan AT, Ang KK. Addition of bevacizumab to standard chemoradiation for locoregionally advanced nasopharyngeal carcinoma (RTOG 0615): a phase 2 multi-institutional trial. Lancet Oncol. 2012 Feb;13(2):172-80. doi: 10.1016/S1470-2045(11)70303-5. Epub 2011 Dec 15. PMID 22178121
- [Result] Liu Z, Wang D, Li G, Yi M, Zhang Z, Zhong G, Xu L, Jiang R, Zheng Y, Huang L, Peng Y, Liang L, Li J, Liu Y, Lai J, Lv X, Xu Y, Liu Q, Wang Z, Liu Z, Yang Q, Nie L, Lei J, Huang X, Liu Z, Jiang W. Neoadjuvant with low-dose radiotherapy, tislelizumab, albumin-bound paclitaxel, and cisplatin for resectable locally advanced head and neck squamous cell carcinoma: phase II single-arm trial. Nat Commun. 2025 May 17;16(1):4608. doi: 10.1038/s41467-025-59865-1. PMID 40382318
- [Result] Wang H, Yao Z, Kang K, Zhou L, Xiu W, Sun J, Xie C, Yu M, Li Y, Zhang Y, Zheng Y, Lin G, Pan X, Wu Y, Luo R, Wang L, Tang M, Liao S, Zhu J, Zhou X, Zhang X, Xu Y, Liu Y, Peng F, Wang J, Xiang L, Yin L, Deng L, Huang M, Gong Y, Zou B, Wang H, Wu L, Yuan Z, Bi N, Fan M, Xu Y, Tong R, Yi L, Gan L, Xue J, Mo X, Chen C, Na F, Lu Y. Preclinical study and phase II trial of adapting low-dose radiotherapy to immunotherapy in small cell lung cancer. Med. 2024 Oct 11;5(10):1237-1254.e9. doi: 10.1016/j.medj.2024.06.002. Epub 2024 Jul 3. PMID 38964333
- [Result] Li S, Li K, Wang K, Yu H, Wang X, Shi M, Liang Z, Yang Z, Hu Y, Li Y, Liu W, Li H, Cheng S, Ye L, Yang Y. Low-dose radiotherapy combined with dual PD-L1 and VEGFA blockade elicits antitumor response in hepatocellular carcinoma mediated by activated intratumoral CD8+ exhausted-like T cells. Nat Commun. 2023 Nov 24;14(1):7709. doi: 10.1038/s41467-023-43462-1. PMID 38001101
- [Result] Chen J, Levy A, Tian AL, Huang X, Cai G, Fidelle M, Rauber C, Ly P, Pizzato E, Sitterle L, Piccinno G, Liu P, Durand S, Mao M, Zhao L, Iebba V, Felchle H, Mallard de La Varende AL, Fischer JC, Thomas S, Greten TF, Jones JC, Monge C, Demaria S, Formenti S, Belluomini L, Dionisi V, Massard C, Blanchard P, Robert C, Quevrin C, Lopes E, Clemenson C, Mondini M, Meziani L, Zhan Y, Zeng C, Cai Q, Morel D, Sun R, Laurent PA, Mangoni M, Di Cataldo V, Arilli C, Trommer M, Wegen S, Neppl S, Riechelmann RP, Camandaroba MP, Neto ES, Fournier PE, Segata N, Holicek P, Galluzzi L, Buque A, Alves Costa Silva C, Derosa L, Kroemer G, Chen C, Zitvogel L, Deutsch E. Low-dose irradiation of the gut improves the efficacy of PD-L1 blockade in metastatic cancer patients. Cancer Cell. 2025 Mar 10;43(3):361-379.e10. doi: 10.1016/j.ccell.2025.02.010. PMID 40068595
- [Result] Herrera FG, Ronet C, Ochoa de Olza M, Barras D, Crespo I, Andreatta M, Corria-Osorio J, Spill A, Benedetti F, Genolet R, Orcurto A, Imbimbo M, Ghisoni E, Navarro Rodrigo B, Berthold DR, Sarivalasis A, Zaman K, Duran R, Dromain C, Prior J, Schaefer N, Bourhis J, Dimopoulou G, Tsourti Z, Messemaker M, Smith T, Warren SE, Foukas P, Rusakiewicz S, Pittet MJ, Zimmermann S, Sempoux C, Dafni U, Harari A, Kandalaft LE, Carmona SJ, Dangaj Laniti D, Irving M, Coukos G. Low-Dose Radiotherapy Reverses Tumor Immune Desertification and Resistance to Immunotherapy. Cancer Discov. 2022 Jan;12(1):108-133. doi: 10.1158/2159-8290.CD-21-0003. Epub 2021 Sep 3. PMID 34479871
- [Result] Zhou L, Liu Y, Wu Y, Yang X, Spring Kong FM, Lu Y, Xue J. Low-dose radiation therapy mobilizes antitumor immunity: New findings and future perspectives. Int J Cancer. 2024 Apr 1;154(7):1143-1157. doi: 10.1002/ijc.34801. Epub 2023 Dec 7. PMID 38059788
- [Result] Herrera FG, Romero P, Coukos G. Lighting up the tumor fire with low-dose irradiation. Trends Immunol. 2022 Mar;43(3):173-179. doi: 10.1016/j.it.2022.01.006. Epub 2022 Jan 31. PMID 35105519
- [Result] Zhang Z, Liu X, Chen D, Yu J. Radiotherapy combined with immunotherapy: the dawn of cancer treatment. Signal Transduct Target Ther. 2022 Jul 29;7(1):258. doi: 10.1038/s41392-022-01102-y. PMID 35906199
- [Result] Yang Y, Pan J, Wang H, Zhao Y, Qu S, Chen N, Chen X, Sun Y, He X, Hu C, Lin L, Yu Q, Wang S, Wang G, Lei F, Wen J, Yang K, Lin Z, Guo Y, Chen S, Huang X, Wu Y, Liang L, Chen C, Bai F, Ma X, Zhang Y, Leaw S, Zhang L, Fang W. Tislelizumab plus chemotherapy as first-line treatment for recurrent or metastatic nasopharyngeal cancer: A multicenter phase 3 trial (RATIONALE-309). Cancer Cell. 2023 Jun 12;41(6):1061-1072.e4. doi: 10.1016/j.ccell.2023.04.014. Epub 2023 May 18. PMID 37207654
- [Result] Yang Y, Qu S, Li J, Hu C, Xu M, Li W, Zhou T, Shen L, Wu H, Lang J, Hu G, Luo Z, Fu Z, Qu S, Feng W, Chen X, Lin S, Zhang W, Li X, Sun Y, Lin Z, Lin Q, Lei F, Long J, Hong J, Huang X, Zeng L, Wang P, He X, Zhang B, Yang Q, Zhang X, Zou J, Fang W, Zhang L. Camrelizumab versus placebo in combination with gemcitabine and cisplatin as first-line treatment for recurrent or metastatic nasopharyngeal carcinoma (CAPTAIN-1st): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2021 Aug;22(8):1162-1174. doi: 10.1016/S1470-2045(21)00302-8. Epub 2021 Jun 23. PMID 34174189
- [Result] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi YR, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Liu Z, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Feng H, Yao S, Keegan P, Xu RH. Toripalimab or placebo plus chemotherapy as first-line treatment in advanced nasopharyngeal carcinoma: a multicenter randomized phase 3 trial. Nat Med. 2021 Sep;27(9):1536-1543. doi: 10.1038/s41591-021-01444-0. Epub 2021 Aug 2. PMID 34341578
- [Result] Prawira A, Oosting SF, Chen TW, Delos Santos KA, Saluja R, Wang L, Siu LL, Chan KKW, Hansen AR. Systemic therapies for recurrent or metastatic nasopharyngeal carcinoma: a systematic review. Br J Cancer. 2017 Dec 5;117(12):1743-1752. doi: 10.1038/bjc.2017.357. Epub 2017 Oct 24. PMID 29065104
- [Result] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Result] Chen YP, Chan ATC, Le QT, Blanchard P, Sun Y, Ma J. Nasopharyngeal carcinoma. Lancet. 2019 Jul 6;394(10192):64-80. doi: 10.1016/S0140-6736(19)30956-0. Epub 2019 Jun 6. PMID 31178151